CLINICAL TRIAL: NCT03749421
Title: Prospective Study of the Prosigna Assay on Neoadjuvant Clinical Decision-making in Women With HR+/Her2- Breast Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: NanoString Technologies, Inc. (Industry)
Responsible Party: Principal Investigator, Sara Tolaney, MD, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 18-281
Record Dates: First submitted 2018-10-19; First posted 2018-11-21 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prosigna Assay: * Biopsy specimen will be subject to molecular profiling via the Prosigna PAM-50 assay
  * The results of Prosigna assay will be provided to the study team in a standardized report.
  * This report will include the patient's intrinsic subtype, ROR score, and general risk (high, intermediate, low).
  Interventions: Other: Prosigna PAM-50 assay

INTERVENTIONS:
Other: Prosigna PAM-50 assay — Looks at the gene activity of a person's cancer cells to determine the likely outcome or course of a disease (prognosis) and predict the benefit of chemotherapy or endocrine therapy after breast surgery

SUMMARY:
This research study is evaluating a genomic analysis called Predictor Analysis of Microarray 50 (PAM50, by Prosigna®) as a tool to possibly guide the participant and the treating physician to choose the most personalized pre-operative treatment for breast cancer.

DETAILED DESCRIPTION:
As the investigators understanding of how ER-positive breast cancer (a type of cancer in which the cells need the hormone estrogen to grow) improves, more treatment decisions are being tailored to an individual's unique genetic makeup. National medical guidelines now include the routine use of tumor profiling tests, like the Prosigna® assay, which look at the gene activity of a person's cancer cells to determine the likely outcome or course of a disease (prognosis) and predict the benefit of chemotherapy or endocrine therapy after breast surgery.

Currently, the Prosigna® assay (also called PAM-50) is FDA approved as a tool that physicians can use to help make decisions about a patient's treatment after their breast surgery. In these cases, physicians run this test using tumor tissue from a patient's breast surgery. However, the Prosigna® assay is not approved for use preoperatively, or before surgery.

Previous studies showed that the Prosigna® assay was able to identify tumor types that were more likely to benefit from treatment before surgery (whether it's hormonal therapy or chemotherapy). In this study, the investigators will use tumor tissue from the participant's biopsy to run the Prosigna® assay. The test may give both the participant and the investigators more information about the best possible treatment option for the participant before surgery.

This study is being done to determine how Prosigna® assay results may affect the physician's choice of treatment before surgery and how well patients understand the test and its implications.

ELIGIBILITY:
Inclusion Criteria:

* Patients pre- or post-menopausal must have histologically confirmed early stage/locally advanced invasive breast cancer
* ER or PR ≥ 1% by immunohistochemistry (IHC)
* HER2-negative status, according to guidelines by ASCO CAP guidelines:

https://www.asco.org/practice-guidelines/quality-guidelines/guidelines/breast-cancer#/9751

* Tumor size ≥ 0.5cm (clinical or radiographic measurements)
* Any nodal status allowed
* Age > 18 years old
* Felt to be a possible candidate for neoadjuvant systemic therapy by their treating physician

Exclusion Criteria:

* ER-negative and PR-negative invasive breast cancer (< 1% by IHC)
* Known metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are considered possible candidates for neoadjuvant treatment, irrespective whether chemotherapy or endocrine therapy, by clinical-pathologic features.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The extent to which the Prosigna test results will change physician's pre-test decision regarding neoadjuvant treatment of patients with stage II-III ER/PR+, HER2-negative breast cancer | 2 years
  Questionnaires will be used to record neoadjuvant treatment decisions pre- and post-test. Data will be summarized in a contingency table, and the extent to which decisions changed will be estimated as the proportion of discordant responses and reported with a two-sided exact 95% confidence interval.

SECONDARY OUTCOMES:
The association of pCR/RCB following neoadjuvant therapy with Risk of recurrence (ROR). | 2 years
  The association of the Prosigna test results to pathologic outcomes will be explored marginally in all patients who receive neoadjuvant treatment, and non-parametric Wilcoxon rank sum and Spearman test of correlation with two-sided alpha = 0.05 will be used to make inferences. Non-linear spline regression techniques will be used to explore the relationship between pre-treatment molecular phenotypes of response to neoadjuvant treatment.
To assess if treatment change was based on ROR score, intrinsic subtype or both | 2 years
  Non-linear spline regression techniques will be used to explore the relationship between pre-treatment molecular phenotypes and response to neoadjuvant treatment. On the "Post-Prosigna Physician Questionnaire" physicians will be asked which of these item (ROR score, instrinsic subtype, or both) contributed to their neoadjuvant treatment decision-making.
To evaluate physicians' confidence in their therapy before and after the test | 2 years
  Physicians will complete pre-test and post-test questionnaires that measure their confidence at each timepoint. The pre-test questionnaire will examine the percentage of physicians who are confident about their treatment recommendation. The same questions about confidence in diagnosis and treatment will be realized after Prosigna results and rates will be compared.
To evaluate patients' confidence in their therapy before and after the test | 2 years
  Patients will complete pre-test and post-test questionnaires to measure their confidence at each timepoint. The pre-test questionnaire will examine the percentage of patients who understand their diagnosis and how Prosigna works and who are confident in treatment recommendation. The same question about diagnosis and treatment will be realized after Prosigna results and rates will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tolaney, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Corti C, Chu X, Exman P, Kline DM, Priedigkeit NM, Mayer EL, Waks AG, Hughes ME, Abravanel DL, Giordano A, Curigliano G, Lin NU, King TA, Jeselsohn RM, Manning DK, Dillon DA, Mittendorf EA, Tayob N, Tolaney SM. Impact of the Prosigna assay on neoadjuvant treatment decision-making in patients with early-stage HR-positive/HER2-negative breast cancer: a single-center prospective observational study. ESMO Open. 2025 Aug;10(8):105521. doi: 10.1016/j.esmoop.2025.105521. Epub 2025 Jul 25. PMID 40714511